CLINICAL TRIAL: NCT02267135
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Demonstrate the Efficacy of Subcutaneous Secukinumab [300 mg] as Assessed by the Psoriasis Scalp Severity Index (PSSI) at 12 Weeks of Treatment, Compared to Placebo, and to Assess Safety and Tolerability up to 24 Weeks in Adult Subjects With Moderate to Severe Scalp Psoriasis
Brief Title: Efficacy and Safety of Subcutaneous Secukinumab in Adults With Moderate to Severe Scalp Psoriasis
Acronym: SCALP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457AUS01
Record Dates: First submitted 2014-09-30; First posted 2014-10-17 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Scalp Psoriasis
Keywords: scalp psoriasis, plaque psoriasis, secukinumab, AIN457, biologic, monoclonal antibody, psoriasis, AIN457A
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secukinumab (Experimental): Eligible patients will receive secukinumab 300 mg once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by monthly dosing starting at Week 8 through Week 20 inclusive
  Interventions: Biological: Secukinumab 300 mg
- Placebo (Placebo Comparator): Eligible patients will receive placebo doses once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by a dose after four weeks at Week 8. Prior to taking the Week 12 dose, the patient will be assessed for response to treatment using the Psoriasis Scalp Severity Index (PSSI). If the subject is a responder, the subject will continue on placebo dosing weekly at Weeks 12, 13, 14, 15 and 16 and then after four weeks at Week 20. Subjects who are not responders will be switched to treatment with secukinumab 300 mg and will dose once weekly at Weeks 12, 13, 14, 15 and 16 and then after four weeks at Week 20.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab 300 mg — Secukinumab 300 mg will be provided in 1 mL prefilled syringes of 150 mg. Each dose of 300 mg secukinumab will consist of two secukinumab 150 mg injections once weekly for 5 weeks (Baseline, Weeks 1, 2, 3 and 4), followed by dosing every four weeks starting at Week 8 through Week 20 inclusive. In order to maintain the blinding, patients will receive additional placebo injections at Weeks 13, 14 and 15. The patients (or caregivers) will self-inject each dose at the study site under the supervision of site personnel when injections occur of days of study visits. The injections not occurring during a study visit will be done by the patients (or caregivers) at home.
  Other Names: AIN457 300 mg
  Arms: Secukinumab
Biological: Placebo — Placebo will be provided in 1 mL prefilled syringe. Each placebo dose will consist of two placebo injections once weekly for five weeks (Baseline, Weeks 1, 2, 3 and 4), then after four weeks at Week 8. At Week 12, PSSI responders will continue on placebo and receive their injections once weekly for five weeks (Weeks 12, 13, 14, 15 and 16), then followed by dosing after four weeks at Week 20. PSSI non-responders will be switched to receive 300 mg secukinumab at Weeks 12, 13, 14, 15 and 16, then after four weeks at Week 20. The patients (or caregivers) will self-inject each dose at the study site under the supervision of site personnel when injections occur on days of study visits. The injections not occurring during a study visit will be done by the patients (or caregivers) at home.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of secukinumab compared to placebo in adult patients who have moderate to severe scalp psoriasis that is poorly controlled by current psoriasis treatments.

ELIGIBILITY:
Inclusion Criteria:

* Chronic scalp psoriasis for at least the previous six months
* Moderate to severe scalp psoriasis as defined by a PSSI score of ≥12 and 30% or higher of scalp surface area affected
* Must be candidates for systemic therapy, which means having scalp psoriasis inadequately controlled by topical treatments (corticosteroids), and/or phototherapy, and/or previous systemic therapy.

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque
* Drug-induced psoriasis (e.g., new onset or current exacerbation from β-blockers, calcium channel inhibitors)
* Ongoing use of prohibited treatments (e.g., topical or systemic corticosteroids, UV therapy)
* Prior exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL17A or IL-17RA receptors
* Use of other investigational drugs within 30 days prior to study entry, or within a period of 5 half-lives of the investigational treatment, whichever is longer
* Active, ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of secukinumab
* Active system infections (with the exception of the common cold) during the two weeks prior to starting study treatment
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis
Locations (16):
- United States (16):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Andover, Massachusetts
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Gahanna, Ohio
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=38

RESULTS

PARTICIPANT FLOW:
Groups:
- Secukinumab: Eligible patients received secukinumab 300 mg once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by monthly dosing starting at Week 8 through Week 20 inclusive
- Placebo: Eligible participants received placebo doses once weekly at Baseline, Weeks 1, 2, 3 and 4 followed by a dose after four weeks at Week 8. Prior to taking the Week 12 dose, participants were assessed for response to treatment using the Psoriasis Scalp Severity Index (PSSI). If the participant was a responder, the participant continued on placebo through Week 20. Participants who were not responders were switched to treatment with secukinumab 300 mg.
Period: Period 1 (Randomized Set)
Arm/Group | Secukinumab | Placebo
Started | 51 | 51
Completed | 50 | 47
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2 (Randomized Set)
Arm/Group | Secukinumab | Placebo
Started | 50 | 47
Completed | 46 | 46
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Customized [Mean (Standard Deviation); unit: Age (years)]
  Mean | 42.7 (13.39) [19 to 68] | 41.1 (14.17) [18 to 69] | 41.9 (13.74) [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 27 | 21 | 48

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Scalp Severity Index 90 (PSSI 90)
Description: PSSI 90 response (yes) at Week 12; PSSI 90 response means at least a 90% improvement in scalp psoriasis
  Percentage of participants with Psoriasis Scalp Severity Index 90 (PSSI 90) response of "yes"
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 52.9 | 2.0
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; adjusted for body weight (< 90 kg, ≥ 90 kg); Difference between percentages = 51, 95% CI 2-sided [37 to 65]

2. Secondary Outcome: Secondary: Investigator's Global Assessment Model 2011 (IGA Mod 2011) Score of 0 or 1 (Scalp Only)
Description: IGA mod 2011 score of 0 or 1 (scalp only) response at Week 12 (non-responder imputation); IGA mod 2011 score of 0 means no sign of scalp psoriasis, and IGA score of 1 means almost no scalp psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 56.9 | 5.9

3. Secondary Outcome: Change From Baseline in PSSI Score
Description: Change from baseline in Psoriasis Scalp Severity Index (PSSI) score. PSSI score ranges from 0-72 with 72 being severe
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Scores on a scale | -25.47 (17.052) | -5.98 (12.868)

4. Secondary Outcome: Psoriasis Scalp Severity Index 75 (PSSI 75) Response
Description: PSSI 75 response (yes) at Week 12 (non-responder imputation); PSSI 75 response means at least a 75% improvement in scalp psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 62.7 | 5.9

5. Secondary Outcome: Psoriasis Scalp Severity Index 100 (PSSI 100) Response
Description: PSSI 100 response (yes) at Week 12 (non-responder imputation); PSSI 100 response means no sign of scalp psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 35.3 | 0.0

6. Secondary Outcome: Time to 50% Reduction in PSSI Score up to Week 12
Description: Time to 50% reduction in PSSI score up to week 12 was estimated for drug arm
  The median time to reduction was not estimable for placebo because a 50% reduction in PSSI score was not achieved by enough participants receiving placebo
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Secukinumab
Number analyzed (Participants) | 51
weeks | 3.29 [2.43 to 8.14]

7. Secondary Outcome: Psoriasis Area and Severity Index 75 (PASI 75)
Description: PASI 75 response (yes) at Week 12 (non-responder imputation); PASI 75 response means at least a 75% improvement in body psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of participants | 64.7 | 2.0

8. Secondary Outcome: Psoriasis Area and Severity Index 90 (PASI 90)
Description: PASI 90 response (yes) at Week 12 (non-responder imputation); PASI 90 response means at least a 90% improvement in body psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 47.1 | 0.0

9. Secondary Outcome: Psoriasis Area and Severity Index 100 (PASI 100)
Description: PASI 100 response (yes) at Week 12 (non-responder imputation); PASI 100 response means no sign of body psoriasis
Time Frame: 12 weeks
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 23.5 | 0.0

10. Secondary Outcome: Investigator's Global Assessment Model 2011 (GA Mod 2011) Score of 0 or 1 (Entire Body Including Scalp)
Description: IGA mod 2011 score of 0 or 1 (entire body including scalp); IGA mod 2011 score of 0 means no sign of psoriasis, and IGA mod 2011 score of 1 means almost no psoriasis
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Number; unit: Percent of Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Percent of Participants | 52.9 | 3.9

11. Secondary Outcome: Change From Baseline in Subject Assessment of Pain
Description: Change from baseline in the Subject Assessment of Pain
  Scale of 0-10 with 10 being the most painful
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Scores on a scale | -1.43 (3.233) | 1.04 (2.615)

12. Secondary Outcome: Change From Baseline in Subject Assessment of Itching
Description: Change from baseline in the Subject Assessment of Itching
  Scale of 0-10 with 10 being the most itchy
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Scores on a scale | -4.10 (3.008) | -0.24 (2.840)

13. Secondary Outcome: Change From Baseline in Subject Assessment of Scaling (Scalp Only)
Description: Change from baseline in the Subject Assessment of Scaling (scalp only)
  Scale of 0-10 with 10 being the most scaling
Time Frame: 12 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 51 | 51
Scores on a scale | -5.24 (2.861) | -0.65 (2.763)

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Treatment Period 1 Secukinumab 300 mg: Treatment Period 1 Secukinumab 300 mg
- Treatment Period 1 Placebo: Treatment Period 1 Placebo
- Treatment Period 2 Placebo/Secukinumab 300 mg: Treatment Period 2 Placebo/Secukinumab 300 mg
Arm/Group | Treatment Period 1 Secukinumab 300 mg | Treatment Period 1 Placebo | Treatment Period 2 Placebo/Secukinumab 300 mg | Treatment Period 1 & 2: Any Secukinumab
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/51 | 1/46 | 1/96
Other Adverse Events (participants affected / at risk) | 8/51 | 5/51 | 5/46 | 5/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1 Secukinumab 300 mg (N=51) | Treatment Period 1 Placebo (N=51) | Treatment Period 2 Placebo/Secukinumab 300 mg (N=46) | Treatment Period 1 & 2: Any Secukinumab (N=96)
CELLULITIS (Infections and infestations) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period 1 Secukinumab 300 mg (N=51) | Treatment Period 1 Placebo (N=51) | Treatment Period 2 Placebo/Secukinumab 300 mg (N=46) | Treatment Period 1 & 2: Any Secukinumab (N=96)
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 3 | 3
NASOPHARYNGITIS (Infections and infestations) | 3 | 1 | 1 | 1
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e., data from all sites) in the clinical trial.